CLINICAL TRIAL: NCT07060703
Title: Clinical and Paraclinical Characterization of Osseous Anomalies of the Long Bones of Patients With Klippel Trénaunay Syndrome
Acronym: KTSOS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-A02765-40
Record Dates: First submitted 2024-09-12; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-03

CONDITIONS: Radiological Bone Phenotype Description of Patients With KTS ( Klippel-Trénaunay Syndrome )

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiological Bone Phenotype Description of Patients With KTS (Other)
  Interventions: Diagnostic Test: Osteodensitometry

INTERVENTIONS:
Diagnostic Test: Osteodensitometry — exploration of long bones using non-invasive Guided Wave Velocity (GWV) technology.
  comparison of ultrasound parameters (cortical thickness and porosity, among others) with BMD values (spine, right and left femoral necks) obtained by DXA.
  [Time Frame: 20 MIN]
  Other Names: non-invasive technology Speed of Guided Waves

SUMMARY:
Clinical and paraclinical characterization of osseous anomalies of the long bones of patients with Klippel Trénaunay syndrome

DETAILED DESCRIPTION:
The objective is to better characterize bone damage in KTS as well as their risks in the shorter or medium term (potentially higher risks of long bone fractures, hemorrhagic risks in the event of a long bone fracture, osteoarthritis risks or risk osteoporosis) as well as the need for rheumatological care in the care pathway.

ELIGIBILITY:
Inclusion Criteria:

Vascular malformation such as Klippel-Trénaunay syndrome or Capillary malformations (CM) + venous malformations (VM) +/- Lymphatic malformations (LM) + limb overgrowth according to ISSVA (International Society for the Study of Vascular Anomalies) classification.

* Signature of study consent by subject of legal age or by 2 legal guardians for minors Patient affiliated to a social security scheme or beneficiary of such a scheme
* Age greater than or equal to 7 years

Exclusion Criteria:

Pregnant or breast-feeding woman Protected person

-

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Quantification of limb-length asymmetry on lower-limb telemetry (absolute values, in mm) compared with the contralateral side | 20 minutes
  The assessment of bone damage includes an X-ray of a weight-bearing pelvis and limb telemetry to detect any limb length abnormalities.

SECONDARY OUTCOMES:
description vascular of the KTS. | 30 MINUTES
  classification of vascular dysplasia using the International Classification of Vascular Anomalies (ISSVA), Hamburg classification, presence or absence of lymphatic involvement, presence or absence of localized or diffuse intravascular coagulopathy, vascular infiltrative bone involvement on MRI.
measurement of bone density (BMD) in the spine and femoral necks, with calculation of the FRAX index. | 20 MINUTES
  quantitative analysis with measurement of bone density (BMD) in the spine and 2 femoral necks by bone densitometry, images obtained by two-photon X-ray absorptiometry or DXA combined with clinical risk factors using the FRAX tool.
exploration of long bones using non-invasive Guided Wave Velocity (GWV) technology. | 20 MINUTES
  comparison of ultrasound parameters (cortical thickness and porosity, among others) with BMD values (spine, right and left femoral necks) obtained by DXA.
description vascular of the KTS. | 20 minutes
  Cortical thickness (Ct.Th) expressed en mm and porosity (Ct.Po) expressed in percentage %.

CONTACTS AND LOCATIONS:
Overall Officials: SOPHIE M BLAISE, INVESTOGATOR, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Chu Grenoble Alpes, La Tronche, France

IPD SHARING:
Plan to Share IPD: No